CLINICAL TRIAL: NCT07145814
Title: Dexmedetomidine Dose-Dependent Modulation of Lung Function and AQP1 Expression During One-Lung Ventilation in Adults Undergoing Thoracoscopic Surgery: A Randomized Controlled Trial
Brief Title: Dexmedetomidine Dose-Dependent on Lung Function and AQP1 in One-Lung Ventilation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Yuanqiang Li, Professor, People's Hospital of Guangxi Zhuang Autonomous Region
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016NXSYYEC-007
Record Dates: First submitted 2025-08-12; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Acute Lung Injury(ALI)
Keywords: Dexmedetomidine; Aquaporins; Lung Function; One-lung ventilation
MeSH Terms: conditions — Acute Lung Injury | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Placebo group received an equivalent volume of 0.9% saline.
  Interventions: Drug: 0.9 % saline
- dexmedetomidine Low Dose group (Experimental): Following Anesthesia induction, dexmedetomidine (DEX) Low Dose group received a DEX loading dose (0.5 µg/kg over 10 min), followed by continuous infusions of 0.3 µg/kg/h, respectively, until 30 minutes before the end of the operation.
  Interventions: Drug: dexmedetomidine 0.3 µg/kg/h
- dexmedetomidine high dose group (Experimental): Following Anesthesia induction, dexmedetomidine (DEX) high dose group received a DEX loading dose (0.5 µg/kg over 10 min), followed by continuous infusions of 0.5 µg/kg/h, respectively, until 30 minutes before the end of the operation.
  Interventions: Drug: dexmedetomidine 0.5 µg/kg/h

INTERVENTIONS:
Drug: dexmedetomidine 0.3 µg/kg/h — Following Anesthesia induction, dexmedetomidine (DEX) Low Dose group received a DEX loading dose (0.5 µg/kg over 10 min), followed by continuous infusions of 0.3 µg/kg/h, respectively, until 30 minutes before the end of the operation.
  Arms: dexmedetomidine Low Dose group
Drug: dexmedetomidine 0.5 µg/kg/h — Following Anesthesia induction, dexmedetomidine (DEX) high dose group received a DEX loading dose (0.5 µg/kg over 10 min), followed by continuous infusions of 0.5 µg/kg/h, respectively, until 30 minutes before the end of the operation.
  Arms: dexmedetomidine high dose group
Drug: 0.9 % saline — Placebo group received an equivalent volume of 0.9% saline.
  Arms: Placebo group

SUMMARY:
This randomized controlled trial evaluated the dose-dependent effects of dexmedetomidine (DEX) on pulmonary function and aquaporin-1 (AQP1) expression during one-lung ventilation (OLV) in thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II
* Age 40-70 years
* Body mass index (BMI) 18-30 kg/m²

Exclusion Criteria:

* Preoperative tumor radiotherapy or chemotherapy
* Immune or endocrine disorders
* Hepatic or renal dysfunction
* Preoperative corticosteroid use
* Recent respiratory infection or chronic lung disease
* Sick sinus syndrome or atrioventricular block
* Preoperative anemia (hemoglobin < 90 g/L)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
aquaporin-1 (AQP1) expression during one-lung ventilation in thoracoscopic surgery | before one-lung ventilation, Immediately after lobectomy
  AQP1 expression, serving as an indicator of pulmonary interstitial water permeability, was assessed by immunohistochemistry (IHC) on lung tissue samples. Two histologically normal specimens (1×1×1 cm³ each) were collected per patient: 1) Before one-lung ventilation: ≥ 5 cm from tumor margin in planned resection area; 2) Immediately after lobectomy: ≥ 5 cm from margin in isolated lung. Tissues were fixed in 10% neutral buffered formalin (24 hours), paraffin-embedded, and sectioned (3 μm). Five random high-power fields (HPF, 400x) per section were evaluated. The percentage of positive cells (0: 0-25%; 1: 26-50%; 2: 51-75%; 3: 76-100%) and staining intensity (0: none; 1: light yellow; 2: brown; 3: dark brown) were scored. The total IHC score (range 0-9) was calculated as (percentage score x intensity score); specimens were classified as low (≤ 4) or high (> 4) AQP1 expression.

SECONDARY OUTCOMES:
Pulmonary function during one-lung ventilation in thoracoscopic surgery, including lung compliance (Cdyn) | pre-dexmedetomidine administration, 60 minutes, 90 minutes, 120 minutes after one-lung ventilation initiation, and 30 minutes after reinstitution of two-lung ventilation
  Radial arterial blood samples were drawn for blood gas analysis at the specified time points. Dynamic lung compliance (Cdyn) was recorded from the anesthesia machine.
Pulmonary function during one-lung ventilation in thoracoscopic surgery, including respiratory index (RI), and oxygenation index (OI). | pre-dexmedetomidine administration, 60 minutes, 90 minutes, 120 minutes after one-lung ventilation initiation, and 30 minutes after reinstitution of two-lung ventilation
  Radial arterial blood samples were drawn for blood gas analysis at the specified time points. The respiratory index (RI) and oxygenation index (OI) were calculated as:
  RI=P(A-aDO2)/PaO2=[(Pb-PH2O) × FiO2-PaO2-PaCO2/RQ]/PaO2. OI= PaO2/FiO2. P(A-aDO2) - alveolar-arterial blood oxygen partial pressure difference, PaCO2 - partial arterial pressure of CO2, Pb - barometric pressure (760 mmHg), pH2O - partial pressure of water vapor (47 mmHg), RQ - respiratory quotient (0.8).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Nanxishan Hospital of Guangxi Zhuang Autonomous Region, Guilin, Guangxi, China

IPD SHARING:
Plan to Share IPD: No